CLINICAL TRIAL: NCT06705959
Title: Can NISS or ISS Better Predict Mortality in Blunt Trauma Patients? A Prospective Study
Brief Title: Comparing NISS and ISS for Mortality Prediction in Trauma Patients
Acronym: ISS/NISS/ER
Status: Recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241122
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Trauma
Keywords: NISS; ISS; Trauma; ER
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this prospective cohort study is to compare the predictive utility of the New Injury Severity Score (NISS) and the Injury Severity Score (ISS) in determining mortality outcomes among trauma patients admitted to emergency rooms (ER) in Iraq.

The main questions it aims to answer are:

* Does the NISS provide a more accurate prediction of mortality than the ISS?
* Are there specific subgroups of trauma patients where one scoring system outperforms the other?

Participants will:

Be assessed using both the NISS and the ISS upon their ER admission. Have their clinical outcomes, including mortality, monitored throughout their hospital stay.

DETAILED DESCRIPTION:
Trauma is a leading global cause of morbidity and mortality, particularly among individuals under 40 years of age, accounting for approximately 5 million deaths annually. To address the challenges of assessing trauma severity, tools like the Injury Severity Score (ISS) and the New Injury Severity Score (NISS) have been developed to predict patient outcomes, including mortality. The ISS, introduced in 1974, is based on the Abbreviated Injury Scale and evaluates the three most severely injured body regions. However, it has limitations, including its inability to account for multiple injuries in the same body region. To overcome these, the NISS was introduced in 1997, summing the squares of the three most severe injuries, irrespective of location, potentially offering improved predictive accuracy in certain trauma populations.

The predictive accuracy of ISS and NISS has been extensively studied, with mixed findings. Meta-analyses and cohort studies suggest both tools are effective, with NISS often demonstrating slightly superior sensitivity and area under the curve (AUC) for mortality prediction. For instance, one analysis reported an AUC of 0.9095 for NISS versus 0.9009 for ISS in predicting mortality. While both tools are considered reliable, NISS's ability to account for multiple severe injuries within the same region makes it particularly advantageous in cases of polytrauma.

Despite these advances, significant heterogeneity exists among studies, largely due to differences in trauma mechanisms, patient populations, and study methodologies. For instance, blunt versus penetrating trauma and age-related factors can influence the tools' performance. Additionally, the lack of standardized reporting and quality assurance in scoring further complicates comparisons, highlighting a need for more uniform research protocols.

In Iraq, where trauma from road traffic accidents and violence is prevalent, evaluating the predictive utility of ISS and NISS is particularly important. Despite the global use of these tools, limited data exists on their effectiveness in Middle Eastern populations, where differences in healthcare infrastructure and injury patterns may affect performance. This study aims to address this gap by comparing the mortality predictive abilities of ISS and NISS in an Iraqi trauma population. Understanding their relative effectiveness in this context could inform better resource allocation, improve trauma care, and guide future research tailored to local needs.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients admitted to the emergency room (ER).
* Patients with documented injury data are sufficient for calculating both the NISS and ISS.
* Patients admitted to the ER within 6 hours of injury.
* Patients providing informed consent (or consent obtained from a legal guardian in cases of incapacity).

Exclusion Criteria:

* Patients under 18 years of age.
* Trauma cases involving burns as the primary injury.
* Patients with incomplete medical records or insufficient data to calculate NISS and ISS.
* Patients with pre-existing terminal conditions (e.g., advanced cancer, end-stage organ failure) unrelated to the trauma.
* Patients who died on arrival or before NISS/ISS assessment could be performed.
* Cases involving pregnant patients, if the primary focus of injury and risk assessment is maternal-fetal outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of trauma patients aged 18 years and older who are admitted to the emergency room (ER) at Al-Kadhimiya Teaching Hospital in Baghdad, Iraq. This group will include individuals with various types of injuries, such as those from road traffic accidents, falls, and assaults, excluding burns as the primary injury.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | In-Hospital Phase (average of 7 days through discharge)
  Mortality (death) during hospitalization
Accuracy Assessment of New Injury Severity Score (NISS) | the first 6 hours after ER admission
  Range: 0 to 75. Higher values indicate worse outcomes, reflecting greater injury severity.
Accuracy Assessment of Injury Severity Score (ISS) | the first 6 hours after ER admission
  Range: 0 to 75 Higher values indicate worse outcomes, reflecting greater injury severity.

SECONDARY OUTCOMES:
Length of Hospitalization | Up to discharge, an average of 7 days
  The total duration of a patient's stay in the hospital, measured from the date of admission to the date of discharge. This includes all days spent in general wards, intensive care units (ICU), and other hospital departments as part of their treatment course.
The requirement for admission to the intensive care unit (ICU) | Up to discharge, an average of 7 days
  The requirement for admission to the intensive care unit (ICU) is determined by the presence of severe clinical deterioration, significant complications, or the need for advanced monitoring and life-support measures.

CONTACTS AND LOCATIONS:
Overall Officials: Anees K Nile, Professor of general surgery, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Palmer CS, Gabbe BJ, Cameron PA. Defining major trauma using the 2008 Abbreviated Injury Scale. Injury. 2016 Jan;47(1):109-15. doi: 10.1016/j.injury.2015.07.003. Epub 2015 Jul 10. PMID 26283084
- [Result] Pape HC, Halvachizadeh S, Leenen L, Velmahos GD, Buckley R, Giannoudis PV. Timing of major fracture care in polytrauma patients - An update on principles, parameters and strategies for 2020. Injury. 2019 Oct;50(10):1656-1670. doi: 10.1016/j.injury.2019.09.021. Epub 2019 Sep 13. PMID 31558277
- [Result] Whitaker IY, Gennari TD, Whitaker AL. The difference between ISS and NISS in a series of trauma patients in Brazil. Annu Proc Assoc Adv Automot Med. 2003;47:301-9. PMID 12941232
- [Result] Hoke MH, Usul E, Ozkan S. Comparison of Trauma Severity Scores (ISS, NISS, RTS, BIG Score, and TRISS) in Multiple Trauma Patients. J Trauma Nurs. 2021 Apr-Jun 01;28(2):100-106. doi: 10.1097/JTN.0000000000000567. PMID 33667204
- [Result] Jamulitrat S, Sangkerd P, Thongpiyapoom S, Na Narong M. A comparison of mortality predictive abilities between NISS and ISS in trauma patients. J Med Assoc Thai. 2001 Oct;84(10):1416-21. PMID 11804251
- [Result] Deng Q, Tang B, Xue C, Liu Y, Liu X, Lv Y, Zhang L. Comparison of the Ability to Predict Mortality between the Injury Severity Score and the New Injury Severity Score: A Meta-Analysis. Int J Environ Res Public Health. 2016 Aug 16;13(8):825. doi: 10.3390/ijerph13080825. PMID 27537902
- [Result] Tohira H, Jacobs I, Mountain D, Gibson N, Yeo A. Systematic review of predictive performance of injury severity scoring tools. Scand J Trauma Resusc Emerg Med. 2012 Sep 10;20:63. doi: 10.1186/1757-7241-20-63. PMID 22964071
- [Result] Rio TGGND, Nogueira LS, Lima FR, Cassiano C, Garcia DFV. Performance of severity indices for admission and mortality of trauma patients in the intensive care unit: a retrospective cohort study. Eur J Med Res. 2023 Dec 4;28(1):559. doi: 10.1186/s40001-023-01532-6. PMID 38049903